CLINICAL TRIAL: NCT02139488
Title: Organ Motion and Early Tumor Response Measurement During Chemotherapy for Esophageal Cancer
Brief Title: Organ Motion and Early Tumor Response Measurement
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: N13OME
Record Dates: First submitted 2014-03-31; First posted 2014-05-15 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Cancer; Chemoradiation
Keywords: Esophageal cancer; Chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fiducial Markers; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- neoadjuvant or definitive chemoradiation: Esophageal cancer patients planned for neoadjuvant or definitive chemoradiation.
  Interventions: Other: Fiducial markers; Other: Fiducial markers, Pet and MRI

INTERVENTIONS:
Other: Fiducial markers
Other: Fiducial markers, Pet and MRI — Insertion of Fiducial markers in esophageal wall.

SUMMARY:
To quantify motion based variation of the target volume of the primary tumor over the course of chemoradiotherapy in esophageal cancer patients, and to use this information to calculate appropriate PTV (planning target volume) margins according to the margins recipe for patients receiving trimodality (neoadjuvant chemoradiation and surgery) or definitive chemoradiation in order to personalize radiation treatment, resulting in either better target coverage or a reduction in normal tissue radiation exposure.

DETAILED DESCRIPTION:
A single center prospective observational study will be performed in esophageal cancer patients. This study registers motion of the esophageal tumor, using 4D planning CT scans and repeated 4D CBCT scanning. Motion of fiducial markers inserted into the esophageal wall, will be used as a surrogate for tumor motion in the limited image quality of CBCT scans.

Patients planned for trimodality treatment will additionally be imaged by serial 4D Pet CT and MRI in week 0 (before start chemoradiotherapy), week 3 (during chemoradiotherapy) and week 10 (just prior to surgery) to observe (early) signs of tumor response.

Patients planned for definitive chemoradiation will not receive extra MRI imaging during treatment because of the inability to correlate this imaging with pathological response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic evidence of invasive adenocarcinoma or squamous cell cancer of the esophagus
2. Patient eligible for trimodality treatment (chemoradiotherapy and surgery) or definitive chemoradiotherapy
3. T3N0M0 or T1-4N1-3M0. Patients with M1 disease solely on the basis of supraclavicular metastasis and not a junction tumor as primary are eligible. (AJCC 7th edition,).
4. WHO performance status ≤2 (WHO scale)
5. Clinically operable for R0 resection in the opinion of an experienced upper gastrointestinal or thoracic surgeon for patients planned for trimodality
6. Tumor localization at least 2cm from the upper esophageal sphincter and invading no more than 5cm into gastric cardia
7. Age ≥ 18 years
8. Written informed consent before endoscopy or EUS

Exclusion criteria:

1. Prior treatment with thoracic surgery or thoracic radiotherapy
2. Pregnancy
3. Severe cardiopulmonary restriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Histologic evidence of invasive adenocarcinoma or squamous cell cancer of the esophagus
  * Patient eligible for trimodality treatment (chemoradiotherapy and surgery) or definitive chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-04-18 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
To quantify motion of the esophageal tumor over the course of chemoradiation | 6 weeks
  The outcome measures will be assessed by tracking the motion of the fiducial markers at the daily 4D CBCT (four dimensional cone beam CT scan). (primary outcome)
  By observing the motion of the fiducial, the exact setup error, breathing motion amplitudes, intra- and inter-fraction motion can be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Francine Voncken, MD, Principal Investigator — NKI-AvL
Locations (1):
- The Netherlands cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
data of two clinic trials will be joined for MRI scans

REFERENCES:
- [Derived] Vollenbrock SE, Voncken FEM, Lambregts DMJ, Maas M, Donswijk ML, Vegt E, Ter Beek LC, van Dieren JM, van Sandick JW, Aleman BMP, Beets-Tan RGH, Bartels-Rutten A. Clinical response assessment on DW-MRI compared with FDG-PET/CT after neoadjuvant chemoradiotherapy in patients with oesophageal cancer. Eur J Nucl Med Mol Imaging. 2021 Jan;48(1):176-185. doi: 10.1007/s00259-020-04917-5. Epub 2020 Jun 22. PMID 32572560